CLINICAL TRIAL: NCT04982575
Title: Efficacy and Safety of Co-administration of Cagrilintide s.c. 2.4 mg and Semaglutide s.c. 2.4 mg Once Weekly in Subjects With Type 2 Diabetes
Brief Title: Research Study to Look at How Well Cagrilintide Together With Semaglutide Works in People With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4862
Record Dates: First submitted 2021-07-16; First posted 2021-07-29 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; cagrilintide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cagrilintide 2.4 mg and semaglutide 2.4 mg (Experimental): Participants will receive cagrilintide and semaglutide once a week as injections for 32 weeks.
  Interventions: Drug: Semaglutide 2.4 mg; Drug: Cagrilintide 2.4 mg
- Cagrilintide 2.4 mg and placebo (semaglutide) (Active Comparator): Participants will receive cagrilintide and placebo (semaglutide) once a week as injections for 32 weeks
  Interventions: Drug: Cagrilintide 2.4 mg; Drug: Placebo (semaglutide)
- Semaglutide 2.4 mg and Placebo (cagrilintide) (Active Comparator): Participants will receive semaglutide and placebo (cagrilintide) once a week as injections for 32 weeks
  Interventions: Drug: Semaglutide 2.4 mg; Drug: Placebo (cagrilintide)

INTERVENTIONS:
Drug: Semaglutide 2.4 mg — Semaglutide administered s.c. (subcutaneously, under the skin) once weekly. Participants will gradually increase the dose until they reach the target dose, and will continue on the this dose once weekly up to 32 weeks
  Arms: Cagrilintide 2.4 mg and semaglutide 2.4 mg; Semaglutide 2.4 mg and Placebo (cagrilintide)
Drug: Cagrilintide 2.4 mg — Cagrilintide administered s.c. (subcutaneously, under the skin) once weekly. Participants will gradually increase the dose until they reach the target dose, and will continue on the this dose once weekly up to 32 weeks
  Arms: Cagrilintide 2.4 mg and placebo (semaglutide); Cagrilintide 2.4 mg and semaglutide 2.4 mg
Drug: Placebo (semaglutide) — Placebo (semaglutide) administered s.c. (subcutaneously, under the skin) once weekly.
  Participants will gradually increase the dose until they reach the target dose, and will continue on the this dose once weekly up to 32 weeks
  Arms: Cagrilintide 2.4 mg and placebo (semaglutide)
Drug: Placebo (cagrilintide) — Placebo (cagrilintide) administered s.c. (subcutaneously, under the skin) once weekly.
  Participants will gradually increase the dose until they reach the target dose, and will continue on the this dose once weekly up to 32 weeks
  Arms: Semaglutide 2.4 mg and Placebo (cagrilintide)

SUMMARY:
This study looks at how well a new medicine called cagrilintide works together with semaglutide on blood sugar levels in people with type 2 diabetes compared to cagrilintide alone or semaglutide alone.

Before a new medicine can be prescribed to people it needs to be tested to see if it is safe and effective.

Participants will either get cagrilintide and semaglutide together or cagrilintide and a dummy medicine or semaglutide and a dummy medicine. Which treatment participants get is decided by chance.

A dummy medicine (placebo) looks like the study medicine but does not contain any active medicine. The dummy medicine is in the study to see if the study medicine works as expected.

Participants will get 2 injections per week on the same day. Participants will take the study medicine with a pen. A pen is a medical tool with a needle used for injections under the skin. The study doctor or staff will show how.

The study will last for about 39 weeks. Participants will have 12 visits at the clinic and 5 phone calls with the study doctor.

At 6 of the clinic visits participants must not eat and drink for 8 hours before the visit (water is allowed).

Women who can become pregnant cannot take part in this study. Only women that are surgically sterilised or post-menopausal are allowed to participate in this study Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period

ELIGIBILITY:
Inclusion Criteria:

* Female of non-childbearing potential or male
* Age above or equal to 18 years at the time of signing informed consent
* Body mass index (BMI) greater than or equal to 27.0 kg/m^2
* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days before screening
* Glycated haemoglobin (HbA1c) of 7.5-10.0% (58-86 mmol/mol) (both inclusive) as assessed by central laboratory at screening
* Stable daily dose(s) ≥ 90 days before screening of the following antidiabetic drug(s) or combination regimen(s) at maximum tolerated or effective dose as judged by the investigator: metformin with or without Sodium-glucose co-transporter-2 (SGLT2) inhibitor

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 days and prior insulin treatment for gestational diabetes are allowed
* Renal impairment with estimated Glomerular Filtration Rate (eGFR) below 60 ml/min/1.73m^2 by central laboratory at screening
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (23):
- United States (23):
  - Uni of Alabama at Birmingham, Birmingham, Alabama
  - Valley Research, Fresno, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - Encompass Clinical Research_Spring Valley, Spring Valley, California
  - New West Physicians,Inc., Golden, Colorado
  - FPA Clinical Research, Kissimmee, Florida
  - Florida Inst For Clin Res, Orlando, Florida
  - Clinical Trial Res Assoc,Inc, Plantation, Florida
  - Ellipsis Group, Alpharetta, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Macoupin Research Group, Gillespie, Illinois
  - MD Medical Research, Oxon Hill, Maryland
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Plains Clinical Research Center, LLC_Fargo, Fargo, North Dakota
  - Holston Medical Group, Kingsport, Tennessee
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Selma Medical Associates, Winchester, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Frias JP, Deenadayalan S, Erichsen L, Knop FK, Lingvay I, Macura S, Mathieu C, Pedersen SD, Davies M. Efficacy and safety of co-administered once-weekly cagrilintide 2.4 mg with once-weekly semaglutide 2.4 mg in type 2 diabetes: a multicentre, randomised, double-blind, active-controlled, phase 2 trial. Lancet. 2023 Aug 26;402(10403):720-730. doi: 10.1016/S0140-6736(23)01163-7. Epub 2023 Jun 23. PMID 37364590

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 17 sites in the United States.
Pre-assignment Details: After randomisation, participants were to continue their pre-trial metformin and sodium-glucose co-transporter-2 (SGLT2) inhibitor background medication throughout the entire trial. The background metformin and SGLT2 inhibitor were to be maintained at the stable, pre-trial dose and at the same frequency during the entire treatment period unless glycaemic rescue treatment was needed or adjustment was required due to safety concerns.
Groups:
- Cagrilintide 2.4 mg + Semaglutide 2.4 mg: Participants received 2.4 milligram (mg) cagrilintide and 2.4 mg semaglutide once-weekly s.c. (subcutaneously, under the skin) injections for 32 weeks. Participants initially received 0.25 mg once weekly and the dose was then escalated once in 4 weeks until the maintenance dose (2.4 mg) was reached: 0.25 mg (week 1 to week 4), 0.5 mg (week 5 to week 8), 1.0 mg (week 9 to week 12), 1.7 mg (week 13 to week 16), 2.4 mg (week 17 to week 32).
- Cagrilintide 2.4 mg + Placebo (Semaglutide): Participants received 2.4 mg cagrilintide and placebo matched to 2.4 mg semaglutide, once-weekly s.c. (subcutaneously, under the skin) injections for 32 weeks. Participants initially received 0.25 mg once weekly and the dose was then escalated once in 4 weeks until the maintenance dose (2.4 mg) was reached: 0.25 mg (week 1 to week 4), 0.5 mg (week 5 to week 8), 1.0 mg (week 9 to week 12), 1.7 mg (week 13 to week 16), 2.4 mg (week 17 to week 32).
- Semaglutide 2.4 mg + Placebo (Cagrilintide): Participants received 2.4 mg semaglutide and placebo matched to 2.4 mg cagrilintide, once-weekly s.c. (subcutaneously, under the skin) injections for 32 weeks. Participants initially received 0.25 mg once weekly and the dose was then escalated once in 4 weeks until the maintenance dose (2.4 mg) was reached: 0.25 mg (week 1 to week 4), 0.5 mg (week 5 to week 8), 1.0 mg (week 9 to week 12), 1.7 mg (week 13 to week 16), 2.4 mg (week 17 to week 32).
Period: Overall Study
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Cagrilintide 2.4 mg + Placebo (Semaglutide) | Semaglutide 2.4 mg + Placebo (Cagrilintide)
Started | 31 | 30 | 31
Completed | 29 | 30 | 29
Not Completed | 2 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analyis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Cagrilintide 2.4 mg + Placebo (Semaglutide) | Semaglutide 2.4 mg + Placebo (Cagrilintide) | Total
Number analyzed (Participants) | 31 | 30 | 31 | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56 (10) | 62 (7) | 57 (10) | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 13 | 33
  Male | 18 | 23 | 18 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 13 | 29
  Not Hispanic or Latino | 21 | 24 | 18 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 5 | 5 | 5 | 15
  White | 26 | 22 | 24 | 72
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin (HbA1c): Cagrilintide 2.4 mg + Semaglutide 2.4 mg Versus Semaglutide 2.4 mg + Placebo (Cagrilintide)
Description: Change in HbA1c from baseline (week 0) to week 32 is presented. The endpoint was evaluated based on the data from in-trial period. The in-trial period is defined as the time interval from date of randomization to date of last contact with trial site. The on-treatment without rescue medication period is a subset of the 'on-treatment' observation period and represents the time period where subjects are considered exposed to trial product but have not initiated any rescue medications.
Time Frame: Week 0, Week 32
Population: Full analysis set included all randomised participants. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Semaglutide 2.4 mg + Placebo (Cagrilintide)
Number analyzed (Participants) | 30 | 30
Percentage of HbA1c
  Change from Baseline - in-trial | -2.2 (0.9) | -1.9 (1.0)
  Change from Baseline - on treatment without rescue | -2.2 (0.9) | -2.0 (1.0)
Statistical Analysis 1: Comparison: Cagrilintide 2.4 mg + Semaglutide 2.4 mg vs Semaglutide 2.4 mg + Placebo (Cagrilintide); The change in HbA1c from baseline was analysed using an ANCOVA (Analysis of Covariance) with randomised treatment and stratification factor as factors and baseline HbA1c as a covariate using retrieved participants multiple imputation of missing data regardless of treatment or stratification; Test type: Other; p = 0.2284, Mixed Models Analysis; Treatment difference = -0.30, 95% CI 2-sided [-0.79 to 0.19]

2. Secondary Outcome: Change in Glycated Haemoglobin (HbA1c): Cagrilintide 2.4 mg + Semaglutide 2.4 mg Versus Cagrilintide 2.4 mg + Placebo (Semaglutide)
Description: Change in HbA1c from baseline (week 0) to week 32 is presented. The endpoint was evaluated based on the data from in-trial period. The in-trial period is defined as the time interval from date of randomization to date of last contact with trial site.
Time Frame: Week 0, Week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Cagrilintide 2.4 mg + Placebo (Semaglutide)
Number analyzed (Participants) | 30 | 30
Percentage point of HbA1c | -2.2 (0.9) | -0.8 (0.9)

3. Secondary Outcome: Percentage Change in Body Weight: Cagrilintide 2.4 mg + Semaglutide 2.4 mg Versus Semaglutide 2.4 mg + Placebo (Cagrilintide)
Description: Percenatge change in body weight from baseline (week 0) to week 32 is presented. The endpoint was evaluated based on the data from in-trial period. The in-trial period is defined as the time interval from date of randomization to date of last contact with trial site.
Time Frame: Week 0, Week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of body weight
Groups:
- Semaglutide 2.4 mg + Placebo (Cagrilintide): Participants received Semaglutide 2.4 mg and 2.4 mg placebo (cagrilintide) once-weekly s.c. (subcutaneously, under the skin) injections for 32 weeks. Participants initially received 0.25 mg once weekly and the dose was then escalated once in 4 weeks until the maintenance dose (2.4 mg) was reached: 0.25 mg (week 1 to week 4), 0.5 mg (week 5 to week 8), 1.0 mg (week 9 to week 12), 1.7 mg (week 13 to week 16), 2.4 mg (week 17 to week 32).
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Semaglutide 2.4 mg + Placebo (Cagrilintide)
Number analyzed (Participants) | 30 | 30
Percentage of body weight | -14.7 (9.3) | -5.0 (4.0)

4. Secondary Outcome: Change in Body Weight (Kilogram): Cagrilintide 2.4 mg + Semaglutide 2.4 mg Versus Semaglutide 2.4 mg + Placebo (Cagrilintide)
Description: Change in body weight from baseline (week 0) to week 32 is presented. The endpoint was evaluated based on the data from in-trial period. The in-trial period is defined as the time interval from date of randomization to date of last contact with trial site.
Time Frame: Week 0, Week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Semaglutide 2.4 mg + Placebo (Cagrilintide)
Number analyzed (Participants) | 30 | 30
Kilogram | -15.4 (10.1) | -5.3 (4.2)

5. Secondary Outcome: Change in Fasting Plasma Glucose (FPG): Cagrilintide 2.4 mg + Semaglutide 2.4 mg Versus Semaglutide 2.4 mg + Placebo (Cagrilintide)
Description: Change in FPG from baseline (week 0) to week 32 is presented. The endpoint was evaluated based on the data from in-trial period. The in-trial period is defined as the time interval from date of randomization to date of last contact with trial site.
Time Frame: Week 0, Week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Semaglutide 2.4 mg + Placebo (Cagrilintide)
Number analyzed (Participants) | 30 | 30
Millimoles per liter (mmol/L) | -3.4 (3.1) | -2.7 (2.3)

6. Secondary Outcome: CGM: Change in Mean Glucose: Cagrilintide 2.4 mg + Semaglutide 2.4 mg Versus Cagrilintide 2.4 mg + Placebo (Semaglutide)
Description: Change in mean glucose from baslline (week 0) to week 32 is presented. The endpoint was evaluated based on the data from in-trial period. The in-trial period is defined as the time interval from date of randomization to date of last contact with trial site.
Time Frame: Week 0, Week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/l)
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Cagrilintide 2.4 mg + Placebo (Semaglutide)
Number analyzed (Participants) | 26 | 28
Millimoles per liter (mmol/l) | -3.5 (2.3) | -1.0 (2.2)

7. Secondary Outcome: Percentage of Time Above Range (TAR) Greater Than 10.0 mmol/L (Greater Than 180 mg/dL) Measured Using CGM (Continuous Glucose Monitoring): Cagrilintide 2.4 mg + Semaglutide 2.4 mg Versus Cagrilintide 2.4 mg + Placebo (Semaglutide)
Description: Percentage of TAR greater than 10.0 mmol/L (greater than 180 mg/dL) at week 32 is presented. The percentage of time spent in glycaemic target range was calculated as 100 times the number of recorded measurements in glycaemic target range greater than 10.0 mmol/L (greater than 180 mg/dL), both inclusive divided by the total number of recorded measurements. The endpoint was evaluated based on the data from in-trial period. The in-trial period is defined as the time interval from date of randomization to date of last contact with trial site.
Time Frame: At week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Cagrilintide 2.4 mg + Placebo (Semaglutide)
Number analyzed (Participants) | 26 | 28
Percentage of time | 10.3 (15.7) | 30.9 (25.2)

8. Secondary Outcome: Percentage of Time in Range (TIR) 3.9-10.0 mmol/L (70-180 mg/dL) Measured Using CGM (Continuous Glucose Monitoring): Cagrilintide 2.4 mg + Semaglutide 2.4 mg Versus Cagrilintide 2.4 mg + Placebo (Semaglutide)
Description: Percentage of TIR 3.9-10.0 mmol/L (70-180 mg/dL) at week 32 is presented. The percentage of time spent in glycaemic target range was calculated as 100 times the number of recorded measurements in glycaemic target range 3.9-10.0 mmol/L (70-180 mg/dL), both inclusive divided by the total number of recorded measurements. The endpoint was evaluated based on the data from in-trial period. The in-trial period is defined as the time interval from date of randomization to date of last contact with trial site.
Time Frame: At week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Cagrilintide 2.4 mg + Placebo (Semaglutide)
Number analyzed (Participants) | 26 | 28
Percentage of time | 88.9 (15.3) | 68.9 (25.1)

9. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial participants administered or using a medicinal product, whether or not considered related to the medicinal product or usage. A TEAE was defined as an event that had onset date (or increase in severity) during the on-treatment observation period. On treatment observation period starts at the date of first dose of trial product and ends at the first date of any of the following; the date of last dose of trial product +35 days for AEs and hypoglycaemic episodes/+ 14 days for other endpoints; the end-date for the 'in-trial' observation period.
Time Frame: From baseline (week 0) to week 37
Population: Safety analysis set included all randomised participants and who take at least 1 dose of trial product.
Measure: Number; unit: Events
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Cagrilintide 2.4 mg + Placebo (Semaglutide) | Semaglutide 2.4 mg + Placebo (Cagrilintide)
Number analyzed (Participants) | 31 | 30 | 31
Events | 21 | 24 | 22

10. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Below 3.0mmol/L (54mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Clinically significant hypoglycaemic episodes (level 2) were defined as episodes that were sufficiently low to indicate serious, clinically important hypoglycaemia with plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL). Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. Number of clinically significant hypoglycaemic episodes (level 2), confirmed by blood glucose (BG) meter or severe hypoglycaemic episodes (level 3) that occurred from week 0 to week 37 are presented. On treatment observation period starts at the date of first dose of trial product and ends at the first date of any of the following; the date of last dose of trial product +35 days for AEs and hypoglycaemic episodes/+ 14 days for other endpoints; the end-date for the 'in-trial' observation period.
Time Frame: From baseline (week 0) to week 37
Population: Safety analysis set included all randomised participants and who take at least 1 dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Cagrilintide 2.4 mg + Placebo (Semaglutide) | Semaglutide 2.4 mg + Placebo (Cagrilintide)
Number analyzed (Participants) | 31 | 30 | 31
Episodes | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline (week 0) to week 37
Description: AEs presented here are TEAEs. TEAE was defined as event that had onset date (or increase in severity) during on-treatment observation period. On treatment observation period starts at date of first dose of trial product & ends at first date of any of following; date of last dose of trial product +35 days for AEs & hypoglycaemic episodes/+ 14 days for other endpoints; end-date for in-trial observation period. SAS included all randomised participants and who take at least 1 dose of trial product.
Arm/Group | Cagrilintide 2.4 mg + Semaglutide 2.4 mg | Cagrilintide 2.4 mg + Placebo (Semaglutide) | Semaglutide 2.4 mg + Placebo (Cagrilintide)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 4/30 | 2/31
Other Adverse Events (participants affected / at risk) | 18/31 | 18/30 | 18/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cagrilintide 2.4 mg + Semaglutide 2.4 mg (N=31) | Cagrilintide 2.4 mg + Placebo (Semaglutide) (N=30) | Semaglutide 2.4 mg + Placebo (Cagrilintide) (N=31)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cagrilintide 2.4 mg + Semaglutide 2.4 mg (N=31) | Cagrilintide 2.4 mg + Placebo (Semaglutide) (N=30) | Semaglutide 2.4 mg + Placebo (Cagrilintide) (N=31)
Acute sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 5 (5) | 5 (5) | 3 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (4) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3)
Fatigue (General disorders) | 3 (3) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (4) | 2 (21) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (10) | 4 (5) | 5 (7)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT04982575/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT04982575/SAP_001.pdf